CLINICAL TRIAL: NCT05085145
Title: The Efficacy of COVID-19 Vaccine in Patients With HIV Infection，a Prospective and Multicenter Clinical Trial
Brief Title: Immunogenicity and Safety of COVID-19 Vaccine in People Living With HIV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ky-2021-7-6-1
Record Dates: First submitted 2021-08-20; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-08

CONDITIONS: People Living With HIV; COVID-19; Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coronavirus vaccination (Experimental): Patients in the experimental need to accept the coronavirus vaccination
  Interventions: Biological: Coronavirus vaccine

INTERVENTIONS:
Biological: Coronavirus vaccine — Coronavirus vaccine was inoculated on day 0 and day 25±3, respectively

SUMMARY:
Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) has caused pandemic since outbreak in 2020. Patients with HIV may be at higher risk than those without HIV for coronavirus disease 2019 (COVID-19). At present, limited data are available on the safety and immunogenicity of coronavirus vaccine for patients with HIV.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, open-label clinical trial. A total of 200 patients with HIV infection were included in this vaccination study. All of the patients will further accept 12 months follow-up study after vaccination. Safety and immunogenicity will be carefully recorded and detected.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years and less than 60 years
2. Patients diagnosed as HIV infection with viral inhibition or preparing to start antivirus therapy were included .
3. The functions of multi-organs were normal or basically normal, and there are no contraindications for vaccination.

Exclusion Criteria:

1. Patients with acute attack of chronic diseases.
2. Patients have history of convulsion, epilepsy, encephalopathy and psychosis.
3. Patients who are allergic to any component of the vaccine, or have a serious history of vaccine allergy.
4. Pregnant or lactating women.
5. Suffering serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, and severe hypertension can not be well controlled by drugs.
6. Patients have severe chronic diseases or diseases can not be controlled well during the progress, such as asthma, diabetes, thyroid disease, etc. Congenital or acquired angioedema / uroedema.
7. Patients who are receiving immunosuppressants such as glucocorticoid.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
The occurence of adverse effects of COVID-19 vaccine in patients with HIV infection | Within 2 months after the first dose of COVID-19 vaccination
  We design a questionnaire for collecting the side effect, answers to the questionnaire are reported and described in a scale of 0-5, where zero indicates the lack of any side effect. Each patient is asked to complete the questionnaire. The questionnaire will be collected on each visit, and blood is drawn for laboratory test.
The immunogenicity and persistence after COVID-19 vaccination in patients with HIV infection | Within 2 months after the first dose of COVID-19 vaccination
  The titers of anti-SARS-CoV-2 antibodies will be detected on each follow-up time for evaluating the efficacy and persistence of COVID-19 vaccine in patients with HIV infection.

SECONDARY OUTCOMES:
The occurence of adverse effects of COVID-19 vaccine in patients with HIV infection | Within 13 months after the first dose of COVID-19 vaccination
  We design a questionnaire for collecting the side effect, answers to the questionnaire are reported and described in a scale of 0-5, where zero indicates the lack of any side effect. Each patient is asked to complete the questionnaire. The questionnaire will be collected on each visit, and blood is drawn for laboratory test.
The immunogenicity and persistence after COVID-19 vaccination in patients with HIV infection | Within 13 months after the first dose of COVID-19 vaccination
  The titers of anti-SARS-CoV-2 antibodies will be detected on each follow-up time for evaluating the efficacy and persistence of COVID-19 vaccine in patients with HIV infection.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-juan Li, MD, Study Director — Beijing 302 Hospital
Locations (1):
- The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No